CLINICAL TRIAL: NCT03541655
Title: A Phase 2, Randomized, Single-Blind, Active-Control, Parallel Group Study to Evaluate Safety and Activity of a Single Administration of F14 for Management of Postoperative Pain in Participants Undergoing Unilateral Total Knee Replacement
Brief Title: Safety and Activity of F14 for Management of Pain Following Total Knee Replacement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arthritis Innovation Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 100-CIP01-P
Record Dates: First submitted 2018-05-08; First posted 2018-05-30 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Total Knee Replacement; Postoperative Pain
Keywords: total knee replacement; pain; celecoxib; intra-articular
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Bupivacaine; Celecoxib

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of care analgesia (Active Comparator): 0.25% Bupivacaine HCl administered following total knee replacement
  Interventions: Drug: Bupivacaine HCl
- F14 (celecoxib) (Experimental): 3.5 mL dose of F14 (celecoxib) concurrent with 0.25% Bupivacaine HCl administered following total knee replacement
  Interventions: Drug: Bupivacaine HCl; Drug: F14 (celecoxib)

INTERVENTIONS:
Drug: Bupivacaine HCl — 0.25% Bupivacaine HCl
  Other Names: Marcaine
Drug: F14 (celecoxib) — Celecoxib in novel drug delivery system (BEPO™)
  Arms: F14 (celecoxib)

SUMMARY:
The safety and activity of a single, 3.5 mL dose of F14 (celecoxib) concurrent with standard of care analgesia administered following total knee replacement will be compared to standard of care analgesia alone.

DETAILED DESCRIPTION:
This is a randomized, single-blind, active control study in participants undergoing primary unilateral total knee replacement (TKR). Fifty (50) participants will be randomized 1:1 to receive either a single, 3.5 mL dose of F14 (celecoxib) concurrent with standard of care analgesia, or only standard of care analgesia. F14 will be administered into the joint space at the end of surgery and just prior to wound closing. Safety will be evaluated through recording of adverse events, vital signs, ECG, physical and knee-specific examinations, laboratory blood tests and standing x-rays of the TKR obtained at 3 and 12 months. Post-operative pain will be assessed using visual analog scores (VAS) and Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaires and the Timed Up and Go test. Concomitant medication usage including MSO4 equivalents will be monitored daily for 3 months with participant drug diaries, and at the 12-month visit. Perceived benefit of analgesia will be compared using the Overall Benefit of Analgesic Score (OBAS). The pharmacokinetic profile of celecoxib in plasma will be assessed up to 3 months. Standardized physical therapy will be implemented post-operatively. Follow-up study visits will occur at 1, 2, 3, 4 (phone) and 6 weeks, 3 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female indicated for primary, unilateral TKR
* Between 45-80 years of age inclusive at the time of signing the informed consent
* Capable of giving signed informed consent and complying with requirements and restrictions listed in the informed consent form (ICF) and in this protocol
* Body Mass Index (BMI) ≤ 40 kg/m²
* Medically stable as determined by the Investigator based on pre-study medical history, physical examination, clinical laboratory tests, and 12-lead electrocardiogram (ECG) findings
* Absence of fixed flexion deformity exceeding 15°
* Absence of varus or valgus deformity exceeding 15°
* Minimum pre-operative flexion arc of 100°
* Absence of steroid, hyaluronic acid, platelet rich plasma, or any other type of therapeutic injection(s) in the index knee within 3 months before scheduled surgery
* American Society of Anesthesiologists Physical Status Classification System (ASA-PSC) score ≤ 3
* Females of childbearing potential with a negative pregnancy test at screening, who agree to employ adequate birth control measures for the full duration of the study
* Has undergone scheduled total knee replacement surgery of the index knee, which in the opinion of the Investigator, will not affect the participant's study follow-up

Exclusion Criteria:

* Allergy or hypersensitivity to active ingredient celecoxib. When an allergy to celecoxib is unknown,allergy or hypersensitivity to sulfonamide antibiotics or sulfa containing drugs
* Active or past infection in the index knee
* Previous total or partial knee arthroplasty in either knee within the past 6 months
* Prior arthroscopy in the index knee in the last 6 months; knee surgery other than arthroscopy (including cruciate ligament, cartilage or osteotomy) in the index knee in the last 12 months; knee surgery in the contralateral knee in the last 12 months (excluding total or partial knee replacement)
* Documented osteonecrosis or arthrotomy within previous 12 months
* Prior or current presence of hardware in index knee other than screws from previous ligament repair that do not require manipulation or removal for TKR surgery
* Other planned major surgery within 12 months of scheduled surgery
* Concurrent painful physical condition that may require analgesic treatment (such as an NSAID or opioid) in the postsurgical period for pain that is not strictly related to the TKR surgery emanating from other lower body joints in the ipsilateral (hip, ankle) or contralateral (hip, knee, ankle) or back (by body diagram)
* Current or historical evidence of any clinically significant disease or condition, especially cardiovascular, pulmonary or neurological conditions that, in the opinion of the Investigator, may increase the risk of surgery or complicate or affect the participant's study follow-up
* Strong narcotic use (e.g. Oxycontin®, Vicodin®, Percocet®) before scheduled study surgery for a prolonged period exceeding 30 days within the last 2 years
* History of alcohol abuse within previous 12 months (score of 4 on CAGE questionnaire)
* Known or suspected history of illicit drug abuse within 1 year before randomization, or history of opioid dependence within 2 years before scheduled surgery (score exceeding 5 on DAST-10 questionnaire)
* Participation in another clinical study involving an investigational product (IP) or device within 30 days before screening or scheduled participation in another clinical study involving an IP or device during the course of this study
* Use of pregabalin or gabapentin, or other drugs for neuropathic pain unless willing to discontinue at least 7 days prior to study surgery
* Current patient-reported seizure disorder
* Current peripheral neuropathy
* Current depression, mood or anxiety disorder (score exceeding 14 on PHQ-9 questionnaire)
* History of complex regional pain syndrome (CRPS)
* Diagnosis of clinically significant liver and/or renal abnormalities within previous 2 years
* Diagnosis of diabetes with HbA1c exceeding 7
* Current inflammatory arthritides (e.g., rheumatoid arthritis, lupus erythematosus, ankylosing spondylitis, psoriatic arthritis), or traumatic bone injuries within 12 months before scheduled surgery, but excepting clinically stable/non-active gout that does not affect the knee and does not interfere with walking
* Treatment with immunosuppressants, antipsychotics, anticholinergics, or anticonvulsants within 1 month of randomization
* Diagnosis of skin disorders including psoriasis, vascular insufficiency ulcers, and chronic venous stasis
* Participants with sleep apnea associated with a history of postoperative delirium. If symptomatic sleep apnea is currently treated with continuous positive airway pressure (CPAP) or bilevel positive airway pressure (BIPAP), use must be continued postoperatively
* History of coronary or vascular stent placed within 3 months (may be extended to 1 year if medically indicated per physician discretion).
* Participation in active or pending personal injury or workers' compensation litigation related to index knee
* Current or planned use of medical marijuana or cannabidiol (CBD), unless willing to discontinue at least 10 days prior to study surgery and for 3 months following study surgery
* Unwilling or unable to discontinue use of NSAIDs within 7 days of scheduled surgery and for 3 months following study surgery, including low-dose aspirin for cardiac prophylaxis
* Has an allergy or contraindication to opioids
* Had a malignancy in the last year, except for non-metastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix
* Positive urine drug screen for disallowed medication at screening or preoperatively on day of study surgery

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Peak pain intensity measured by visual analog scale (VAS) | At 2 weeks
Area under the curve (AUC) of visual analog scale (VAS) pain intensity scores | Through 72 hours
Summed pain intensity difference (SPID) of visual analog scale (VAS) pain intensity scores | Through 72 hours
Functional improvement by Timed Up and Go test | Through 3 months
Total post-surgical opioid consumption (in MSO4 equivalents) | Through 3 months

SECONDARY OUTCOMES:
Peak pain intensity by visual analog score (VAS) | Through 12 months
Pain, stiffness, and physical function by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC Parts A, B, C) | Through 12 months
Time to first rescue medication | Through 3 months
Proportion of participants using rescue medication | Through 3 months
Benefit of analgesia by Overall Benefit of Analgesic Score (OBAS) questionnaire | Through 4 weeks
Celecoxib concentration in plasma | Through 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jared Foran, MD, Principal Investigator — Panorama Orthopedics & Spine Center
Locations (3):
- United States (3):
  - Panorama Orthopedics & Spine Center, Denver, Colorado
  - Midwest Clinical Research Center, Dayton, Ohio
  - Endeavor Clinical Trials, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No